CLINICAL TRIAL: NCT01113398
Title: Phase II Study to Evaluate the Efficacy and Safety of AMG 102 and Avastin in Subjects With Recurrent Malignant Glioma
Brief Title: AMG 102 and Avastin for Recurrent Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Katy Peters (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Katy Peters, Assistant Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00022491
Record Dates: First submitted 2010-04-28; First posted 2010-04-29 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Glioblastoma Multiforme; Gliosarcoma
Keywords: glioblastoma multiforme; gliosarcoma; malignant glioma; glioma; Avastin; bevacizumab; AMG 102; rilotumumab; recurrent; Duke; Pro00022491
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma; Recurrence | interventions — rilotumumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMG 102 with Avastin (Experimental): Avastin will be administered as a continuous intravenous infusion at 10 mg/kg prior to AMG 102, which will be administered as a continuous intravenous infusion by an infusion pump at 20 mg/kg. Subjects will receive infusions every 2 weeks.
  Interventions: Drug: AMG 102; Drug: Avastin

INTERVENTIONS:
Drug: AMG 102 — AMG 102 will be administered as a continuous intravenous infusion by an infusion pump at 20 mg/kg every 2 weeks over 60 or 30 minutes.
  Other Names: rilotumumab
Drug: Avastin — Avastin will be administered as a continuous intravenous infusion at 10 mg/kg every 2 weeks (6-week study cycle) over 60 or 30 minutes. Avastin will be given prior to AMG 102.
  Other Names: Bevacizumab

SUMMARY:
The primary purpose of the study is to assess the response rate of AMG 102 and Avastin treatment in subjects with advanced malignant glioma. Secondary objectives are to estimate overall survival and 6-month progression-free survival rates in this population and to assess the safety of this combination in this population.

Patients must have recurrent histologically confirmed diagnosis of World Health Organization (WHO) grade IV malignant glioma (glioblastoma multiforme or gliosarcoma) with no more than 3 prior progressions. Subjects will receive Avastin and AMG 102 every two weeks. Avastin will be administered prior to AMG 102. Up to 36 adult subjects will take part in this study at Duke.

In initial Phase I and II clinical trials, four potential Avastin-associated safety issues were identified: hypertension, proteinuria, thromboembolic events, and hemorrhage. The most common side effect for AMG 102 have been nausea and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent histologically confirmed diagnosis of WHO grade IV malignant glioma (glioblastoma multiforme or gliosarcoma) with no more than 3 prior progressions.
* Age ≥ 18 years.
* Karnofsky ≥ 60%.
* An interval of at least 4 weeks between either prior tumor biopsy or prior major surgical procedure and study enrollment.
* Bi-dimensionally measurable disease as assessed by magnetic resonance imaging.
* Hemoglobin ≥9.0 g/dl, ANC ≥1500 cells/µl, Platelets ≥125,000 cells/µl (without transfusion within 14 days before enrollment).
* Serum creatinine < 1.5 mg/dl, bilirubin < 1.5 times upper limit of normal, and serum SGOT (AST) and SGPT (ALT) < 2.5 times upper limit of normal.
* For patients on corticosteroids, they must be on a stable dose for 1 week prior to entry, and the dose should not be escalated over entry dose level, if clinically possible.
* Signed informed consent approved by the Institutional Review Board.
* No evidence of active CNS hemorrhage on the baseline MRI or CT scan.
* If sexually active, patients will take contraceptive measures for the duration of treatment as stated in the informed consent.

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Baseline ECG with QTc > 0.45 second
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids.
* Thrombosis or vascular ischemic events within the last twelve months, such as deep venous thrombosis, pulmonary embolism, transient ischemic attack, cerebral infarction, or myocardial infarction.
* Active infection requiring IV antibiotics 7 days before enrollment.
* History of central nervous system bleeding as defined by stroke or intraocular bleed (including embolic stroke) within 6 months before enrollment.
* Evidence of acute intracranial hemorrhage; except for subjects with stable grade 1 hemorrhage.
* Less than 12 weeks from radiation therapy, unless progressive disease outside of the radiation field or 2 consecutive scans or histopathologic confirmation.
* Treated previously with any c-Met or HGF targeted therapy.
* Treated previously with VEGF or VEGFR therapies, including antibodies and tyrosine kinase inhibitors.
* Treated with thalidomide or tamoxifen within 1 week before enrollment unless the patient has recovered from the toxic effects of such therapy.
* Treated with immunotherapeutic agents, vaccines, or MAb therapy within 4 weeks before enrollment unless the patient has recovered from the toxic effects of such therapy.
* Treated with alkylating agents within 4 weeks before enrollment or if the patient has been treated with daily or metronomic chemotherapy unless the patient has recovered from the toxic effects of such therapy.
* Treated with chemotherapy (non-alkylating agents) within 2 weeks before enrollment unless the patient has recovered from the toxic effects of such therapy.
* Less than 4 weeks after surgical resection of the brain tumor or less than 2 weeks after stereotactic biopsy before enrollment unless the patient has recovered from acute side effects of such procedures except for neurological effects.
* Plans to receive surgery, radiation therapy or other elective surgeries during the course of the study.
* Concurrent severe and/or uncontrolled medical disease (e.g. uncontrolled diabetes, congestive cardiac failure, myocardial infarction within 6 months before enrollment) that could compromise participation in the study.
* Concurrent or prior (within 7 days of enrollment) anticoagulation therapy, except: Use of low dose coumadin-type anticoagulants (≤ 2 mg PO QD) low molecular weight heparins (LMWH), e.g. Enoxaparin sodium (Lovenox) and unfractionated heparin for prophylaxis against central venous catheter thrombosis is allowed.
* Grade 2 or greater peripheral edema or effusion (pleural, pericardial, or ascites).
* Inability to comply with study and/or follow-up procedure.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study.

Avastin-Specific Exclusion Criteria

Subjects meeting any of the following criteria are ineligible for study entry:

* Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to Day 1, the day protocol therapy starts.
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Significant vascular disease (e.g. aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) (within 6 months prior to Day 1).
* History of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 28 days prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* Serious, non-healing wound, active ulcer or untreated bone fracture
* Proteinuria as defined by ≥ +1 on urinalysis dipstick
* Known hypersensitivity to any component of Avastin
* Pregnant (positive pregnancy test) or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-08; Primary Completion 2014-11 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine B Peters, MD, PhD, Principal Investigator — Duke University; Mary Lou Affronti, DNP ANP MHSc, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Affronti ML, Jackman JG, McSherry F, Herndon JE 2nd, Massey EC Jr, Lipp E, Desjardins A, Friedman HS, Vlahovic G, Vredenburgh J, Peters KB. Phase II Study to Evaluate the Efficacy and Safety of Rilotumumab and Bevacizumab in Subjects with Recurrent Malignant Glioma. Oncologist. 2018 Aug;23(8):889-e98. doi: 10.1634/theoncologist.2018-0149. Epub 2018 Apr 17. PMID 29666296
- See also: The Preston Robert Tisch Brain Tumor Center — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AMG 102 With Avastin
Started | 36
Completed | 36 (Completed= Discontinued study drug due to disease progression, death, toxicity or any other reason)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AMG 102 With Avastin
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Response
Description: The percentage of participants with a complete or partial response as determined by modified Response Assessment in Neuro-Oncology (RANO) criteria will be determined. Complete Response (CR) is defined as complete disappearance on MR/CT of all enhancing tumor and mass effect, off all corticosteroids (or receiving only adrenal replacement doses) and accompanied by a stable or improving neurologic examination. Partial Response (PR) is defined as greater than or equal to 50% reduction in tumor size on MR/CT by bi-dimensional measurement, on a stable or decreasing dose of corticosteroids and accompanied by a stable or improving neurologic examination. Tumor assessments are done at baseline and the end of every 6-week cycle thereafter.
Time Frame: 2 years
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AMG 102 With Avastin
Number analyzed (Participants) | 36
percentage of participants | 27.8 [15.7 to 44.1]

2. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival is defined as the time in months from the start of protocol treatment until the date of death, or the date of last follow-up if alive. Kaplan-Meier methods will be used to estimate overall survival.
Time Frame: 2 years
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AMG 102 With Avastin
Number analyzed (Participants) | 36
Months | 11.2 [7.0 to 17.5]

3. Secondary Outcome: Six-month Progression-free Survival (PFS6)
Description: The percentage of participants alive and progression-free at 6 months after the start of study treatment will be determined. PFS6 will be calculated from the date study treatment started until the date of progression or death, or the date of last follow-up if participants are alive without progression. Kaplan-Meier methods will be used to estimate survival.
Time Frame: 6 months
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AMG 102 With Avastin
Number analyzed (Participants) | 36
percentage of participants | 41.7 [25.6 to 57.0]

4. Secondary Outcome: Percentage of Participants Who Experience Treatment-related Grade 2 or Greater CNS Hemorrhage or Grade 4 or Greater Non-hematologic Toxicities
Description: The percentage of participants who experience unacceptable toxicity, defined as any treatment-related grade 2 or greater CNS hemorrhage or grade 4 or greater non-hematologic toxicity, will be calculated.
Time Frame: 2 years
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | AMG 102 With Avastin
Number analyzed (Participants) | 36
percentage of participants | 5.5

ADVERSE EVENTS:
Time Frame: From the start of study treatment for a patient until 30 days after treatment is discontinued.
Description: Patients will be evaluated for adverse events (AEs) (all grades), serious AEs, and AEs requiring study drug interruption or discontinuation at each study visit for the duration of their participation in the study. The AEs for this study were collected using CTCAE v.3.0, and have been converted to CTCAE v. 4.0 for entry into ClinicalTrials.gov.
Arm/Group | AMG 102 With Avastin
Serious Adverse Events (participants affected / at risk) | 6/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 102 With Avastin (N=36)
Death NOS (General disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Seizure (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 102 With Avastin (N=36)
Anemia (Blood and lymphatic system disorders) | 6
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 2
Ventricular arrhythmia (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 3
Hearing impaired (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 2
Extraocular muscle paresis (Eye disorders) | 4
Eye disorders - Other, specify (Eye disorders) | 3
Photophobia (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 5
Anal mucositis (Gastrointestinal disorders) | 1
Anal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 3
Fecal incontinence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Gingival pain (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Lip pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Oral hemorrhage (Gastrointestinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 2
Edema face (General disorders) | 2
Edema limbs (General disorders) | 11
Edema trunk (General disorders) | 2
Fatigue (General disorders) | 26
Fever (General disorders) | 1
Gait disturbance (General disorders) | 5
General disorders and administration site conditions - Other, specify (General disorders) | 2
Injection site reaction (General disorders) | 1
Pain (General disorders) | 8
Bronchial infection (Infections and infestations) | 1
Gum infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 5
Lung infection (Infections and infestations) | 2
Mucosal infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Wound infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Burn (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 2
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 3
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 13
Weight gain (Investigations) | 13
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 16
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 18
Hypocalcemia (Metabolism and nutrition disorders) | 19
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 5
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Acoustic nerve disorder NOS (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 4
Cognitive disturbance (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 9
Headache (Nervous system disorders) | 13
Intracranial hemorrhage (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 6
Nervous system disorders - Other, specify (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 5
Seizure (Nervous system disorders) | 12
Tremor (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 5
Confusion (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 10
Proteinuria (Renal and urinary disorders) | 4
Urinary frequency (Renal and urinary disorders) | 5
Urinary incontinence (Renal and urinary disorders) | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 14
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 14
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Purpura (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 7
Skin induration (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 2
Hypertension (Vascular disorders) | 8
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
11/21/14 Amgen notified PI they stopped their own AMG102 studies due to increased risk found in the TX arm on a different study. Dr. Peters decided to stop TX on the 3 current subjects on her study at that time although no increased risks were found.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes